CLINICAL TRIAL: NCT00212628
Title: Controlled Study of ONO-5920 in Patients With Involutional Osteoporosis in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-5920-04; NCT00189865 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Involutional Osteoporosis
Keywords: ONO-5920; osteoporosis; bisphosphonate
MeSH Terms: conditions — Osteoporosis | interventions — YM 529

INTERVENTIONS:
Drug: Minodronic acid hydrate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-5920 in patients with involutional osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who was included in study ONO-5920-02 and completed the medication for two years
2. Other inclusion criteria as specified in the study protocol

Exclusion Criteria:

1. Patients judged to be unsuitable by safety evaluation as clinical trial subjects by the investigator
2. Patients having secondary osteoporosis or another condition that presents low bone mass
3. Other exclusion criteria as specified in the study protocol

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2004-06

PRIMARY OUTCOMES:
New fragility vertebral fracture

SECONDARY OUTCOMES:
New clinical fracture, biochemical markers of bone turnover, height, mean bone mineral density of the lumbar spine (L2-4 BMD), lower back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - Chugoku Region Facility, Chugoku
  - Chubu Region Facility, Chūbu
  - Hokkaido Region Facility, Hokkaido
  - Hokuriku Region Facility, Hokuriku
  - Kanto Region Facility, Kanto
  - Kinki Region Facility, Kinki
  - Kyushu Region Facility, Kyushu
  - Shikoku Region Facility, Shikoku Region Facility
  - Tohoku Region Facility, Tōhoku